CLINICAL TRIAL: NCT00781352
Title: Nitrous Oxide Does Not Increase the Risk of Cancer Recurrence After Colorectal Surgery: A Randomized, Blinded Study
Brief Title: Nitrous Oxide and Risk of Cancer Recurrence After Colorectal Surgery: A Randomized, Blinded Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Edith Fleischmann, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: efno1008
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
Keywords: nitrous oxide; cancer recurrence; colorectal surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nitrous Oxide; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): Colorectal surgery with 65% nitrous oxide administration
  Interventions: Drug: nitrous oxide
- group 2 (Active Comparator): Colorectal surgery with nitrogen administration
  Interventions: Drug: nitrogen

INTERVENTIONS:
Drug: nitrous oxide — 65% nitrous oxide administered during surgery
  Arms: group 1
Drug: nitrogen — Nitrogen administration during surgery
  Arms: group 2

SUMMARY:
This study was developed to test the hypothesis that the risk of colorectal cancer recurrence was similar in patients who were randomly assigned to 65% nitrous oxide or nitrogen during colorectal surgery.

DETAILED DESCRIPTION:
We conducted a 4- to 8-year follow-up of 204 patients with colorectal cancer who were randomly assigned to 65% nitrous oxide (n=97) or nitrogen (n=107), balanced with isoflurane and remifentanil. The primary outcome was the time to cancer recurrence. Our primary analysis was a multivariable Cox-proportional-hazards regression model that included relevant baseline variables. In addition to treatment group, the model considered patient age, tumor grade, dissemination, adjacent organ invasion, vessel invasion, and the number of nodes involved. The study had 80% power to detect a 56% or greater reduction in recurrence rates (i.e., hazard ratio of 0.44 or less) at the 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18-18
* ASA status 1-3
* Informed consent

Exclusion Criteria:

* Acute bowel obstruction
* Minor colon surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 1998-11; Primary Completion 2003-11 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine if the risk of colorectal cancer recurrence was similar in patients who were randomly assigned to 65% nitrous oxide or nitrogen during colorectal surgery. | 270 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Edith Fleischmann, M.D., Principal Investigator — Medical University of Vienna; Daniel I Sessler, M.D., Study Director — The Cleveland Clinic
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fleischmann E, Marschalek C, Schlemitz K, Dalton JE, Gruenberger T, Herbst F, Kurz A, Sessler DI. Nitrous oxide may not increase the risk of cancer recurrence after colorectal surgery: a follow-up of a randomized controlled trial. BMC Anesthesiol. 2009 Feb 3;9:1. doi: 10.1186/1471-2253-9-1. PMID 19192300